CLINICAL TRIAL: NCT00643162
Title: Combination Lexapro and Massage for Treatment in Depression in Older Subjects
Brief Title: Combination Lexapro and Massage for Treatment of Depression in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated recruitment was necessary beyond study capabilities.
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Itai Danovitch, Chairman, Department of Psychiatry, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8648
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Depression
Keywords: Depression; Massage; Lexapro; Alternative Therapy; Anti-depressant
MeSH Terms: conditions — Depression | interventions — Escitalopram; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Swedish Massage (Experimental): Adding massage twice a week, for 8 weeks, and Lexapro in the treatment of depression.
  Interventions: Drug: Lexapro; Behavioral: Massage
- Light-Touch (Sham Comparator): Adding light touch twice a week, for 8 weeks, and Lexapro in the treatment of depression.
  Interventions: Drug: Lexapro; Behavioral: Light touch

INTERVENTIONS:
Drug: Lexapro — 5mg-10mg of lexapro, daily, for 9 weeks for all study participants.
  Other Names: Escitalopram
Behavioral: Light touch — Light touch twice a week, for 8 weeks
  Arms: Light-Touch
Behavioral: Massage — Massage twice a week, for 8 weeks.
  Arms: Swedish Massage

SUMMARY:
Depression is a common and disabling condition which represents a substantial public health concern, especially with the aging of the population in general. In fact, one to four percent of the older population has major depression. Although medication is the main treatment for depression, studies show that only 50% of patients show a significant response to treatment. The response might actually be less in older subjects, and with more adverse side effects due to changes in the metabolism of the older population as well as drug interaction. For these reasons (changes in metabolism and possible drug interactions) the starting dose of the antidepressant Lexapro will be 5mg, instead of 10mg.

To combat the incomplete response to medication, many combined and augmentation strategies have been developed. Examples of this would be an antidepressant medication plus a neuroleptic medication; or an antidepressant medication plus talk therapy. One non-medication treatment that is being considered is massage therapy. Recent data suggest that massage therapy can be useful for the treatment of depression.

This study proposes to perform a controlled trail to assess the effects of massage therapy on symptoms of depression in older subjects with major depression. All of the subjects will receive Lexapro, which is an FDA approved medication for the treatment of depression. Half of the subjects will receive Swedish massage for one hour, twice a week, and the other half will receive light touch for one hour, twice per week for eight weeks. Standardized rating scales that evaluate depression will be used to evaluate the subjects mood.

DETAILED DESCRIPTION:
1. Study Design: This will be an open-label, randomized control trial of concomitant massage therapy and escitalopram pharmacotherapy for the treatment of major depression in the elderly. All subjects who meet inclusion/exclusion criteria will receive escitalopram and also be randomized 1:1 (by computer) to Swedish massage or light touch. Escitalopram (5.0 mg/day, PO) will initially be administered for one week followed by an increase in dose to 10 mg/day for the remainder of the study; Massage or touch will be performed twice per week for 8 weeks. Every effort will be made to have non-consecutive massage/touch visits. The massage group will receive Swedish massage for 50 minutes twice per week. In the "touch" group, the massage therapist will provide gentle touch to the skin in the same distribution as that of the formal Swedish massage for 50 minutes twice per week. Every effort will be made to have one therapist perform all treatments. All assessments will be obtained prior to the first massage each week.
2. Recruitment and Retention: Subjects will be recruited from our outpatient clinic, attendings, as well as by advertising on radio, television, newspaper and our web site.
3. Treatment

   1. Massage: Standard Swedish massage therapy will be employed which includes the systematic manipulation of the soft tissues of the body. It is designed to relax muscles by applying pressure to them against deeper muscles and bones, and rubbing in the same direction as the flow of blood returning to the heart. A routine has been designed whereby the therapist massages different areas of the body in an orderly fashion for specified periods of time. For sham massage (light touch), the massage therapists will provide gentle touch to the skin in the same distribution and duration as that of the formal Swedish massage. As mentioned below, deviations from the structured massage or touch will be recorded in the massage therapist's diary.
   2. Quality control for screening and outcome questionnaires: Kappa co-efficients for diagnostic and inter-rater reliability will be determined at six-month intervals. We routinely maintain kappa values of at >0.85.
4. Outcome Measures: Primary outcome measure for this study will be degree of depression as measured by HAM-D. The secondary outcome measures will include quality of life, HAM-A, Beck Depression Inventory. Raters will be blind to treatment cell and test results.

   Quality control for screening and outcome questionnaires: Kappa co-efficients for diagnostic and inter-rater reliability will be determined at six-month intervals. We routinely maintain kappa values of at >0.85.
5. Statistical Analysis All entries will be blind-verified, and following data entry, results will be checked for obvious outliers and inconsistent values. No single person will have the responsibility for both entry and verification on a given form. Data on computer records will be identifiable by a unique coded identifier to permit matching of records longitudinally. Each record will be logged as it is obtained. An archival record of all data collected, which has passed the above-noted checks, will be maintained on a hard disk. A backup of the archival data will be saved on magnetic tape (DAT tape) and writable CD-ROM archive disks. This copy will be stored in a separate offsite cabinet to ensure the survival of data in case of a natural disaster. A full backup will be made weekly, and stored for at least three months. A CD-ROM backup will be made every three months.

ELIGIBILITY:
Inclusion Criteria:

1. > 60 years of age
2. Unipolar major depression as defined by Structured Clinical Interaction DSM-IV (SCID)
3. HAM-D score of > 17 (21-item scale)]]
4. Not taking antidepressants for at least two weeks, 2 months for fluoxetine and MAOIs]]
5. Capable of giving informed consent.

Exclusion Criteria:

1. Unable to provide informed consent (e.g. severe cognitive impairment)
2. Acute medical condition or exacerbation of chronic medical condition associated with significant distress (pain, protracted fevers, etc.) and requiring active medical treatment.
3. High risk of suicide or violence as assessed by the investigator
4. Current or past history of psychosis or bipolar disorder
5. Use of psychotropic medication and/or psychotherapy outside of the study
6. (Exposure to treatment of fluoxetine or MAOIs in the previous two months; chronic use of benzodiazepine and non-benzodiazepine sedatives, antipsychotics, psychostimulants, mood stabilizing agents, codeine, steroids, anti-inflammatory agents.
7. Alternative medicine use in the preceding 30 days (e.g. acupuncture, herbs, etc.)
8. History of intolerance to massage or contraindication to massage (e.g. skin lesions that prevent direct contact by the therapist)
9. Diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder, schizotypal disorder, psychotic depression or bipolar disorders;
10. MMSE less than 22
11. Alzheimer's Disease Assessment Scale-Cognitive Subscale ³ greater than 12
12. Current drug or alcohol abuse or dependence or history of drug or alcohol abuse or dependence within the past 6 months
13. Unstable medical or neurological conditions that are likely to interfere with the treatment of depression
14. Currently on psychotropic medications including antidepressants or neuroleptics
15. Active suicidal ideation or other safety issues determined by the clinician to not be suitable for inclusion in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itai Danotivtch, Ph.D., M.D., Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center Department of Psychiatry and Behavioral Neurosciences, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 subjects screen failed; 1 subject withdrew consent after screen. Total of 5 subjects were not randomized.
Period: Overall Study
Arm/Group | Swedish Massage | Light-Touch
Started | 7 | 5
Completed | 6 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Swedish Massage | Light-Touch | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Scale (HAM-D) Score
Description: The Hamilton Depression Rating Scale (HAM-D) is a clinician-administered tool used to determine a patient's level of depression before, during, and after treatment. The HAM-D form lists 21 items, but the scoring is based on the first 17 questions. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. The scores from each item are added together to provide a total score. The sum of the scores from the first 17 questions provides an indication for level of depression. 0-7 = normal, 8-13 = mild depression, 14-18 = moderate depression, 19-22=severe depression and ≥ 23=very severe depression.
Time Frame: 9 weeks
Population: A 7th Massage subject completed 6 of 7 visits so his data was carried forward to the final visit. Data from the LT subject who terminated early at Visit 3 was not used. An interim analysis was performed, there was one active subject still in the early stages of the protocol, whose data was not included. The interim analysis became final.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Swedish Massage | Light-Touch
Number analyzed (Participants) | 7 | 3
units on a scale | 13 (7.4) | 10.7 (4.9)
Statistical Analysis 1: Comparison: Swedish Massage vs Light-Touch; Test type: Other; p = .68, t-test, 2 sided; Mean Difference (Final Values) = 2.3, Standard Deviation 6.15

2. Secondary Outcome: Change in Beck Depression Inventory Score
Description: The Beck Depression Inventory (BDI) is a series of 21-question, self-report rating inventory developed at a 5th grade reading level that measures characteristic attitudes and symptoms of depression. It was develop to detect, assess and monitor changes in depressive symptoms. For people who have been clinically diagnosed with depression, scores from 0 to 9 represent minimal depressive symptoms, scores of 10 to 16 indicate mild depression, scores of 17 to 29 indicate moderate depression, and scores of 30 to 63 indicate severe depression.
Time Frame: 9 weeks
Population: Data was not abstracted since interim analysis recommended study closure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Swedish Massage | Light-Touch
Number analyzed (Participants) | 7 | 3
units on a scale | 8.7 (6.6) | 6.3 (6.3)

3. Secondary Outcome: Change in Hamilton Anxiety Scale (HAM-A) Score
Description: The Hamilton Depression Rating Scale (HAM-D) is a clinician-administered tool used to determine a patient's level of anxiety before, during, and after treatment. The HAM-A is a 14-item assessment and each item is scored on a 5-point scale, ranging from 0 = not present to 4 = very severe. The sum of the scores is: 0-17 = mild anxiety, 18-24 = moderate anxiety, 25-30 = severe anxiety, and >30 = very severe anxiety.
Time Frame: 9 weeks
Population: Data was not abstracted since interim analysis recommended study closure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Swedish Massage | Light-Touch
Number analyzed (Participants) | 7 | 3
units on a scale | 5.3 (5.8) | 2.7 (13.1)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Swedish Massage | Light-Touch
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 1/7 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Swedish Massage (N=7) | Light-Touch (N=5)
Cold Symptoms (General disorders) | 1 (1) | 0 (0) — After 2 weeks of taking Lexapro, subject reported symptoms of coughing, sneezing, feeling feverish, fatigue and dizziness and attributed it to a lingering coldAlthough symptoms are not associated with Lexapro, Investigator wanted to report as an AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes